CLINICAL TRIAL: NCT06196762
Title: A Phase 1, First-in-human (FIH),Dose-escalation and Dose-expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of XKH002 in Patients With Advanced or Metastatic Solid Tumors
Brief Title: Phase I of XKH002 Injection in Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Kanova Biopharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XKH002-101
Record Dates: First submitted 2023-11-10; First posted 2024-01-09 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2023-10

CONDITIONS: Advanced or Metastatic Solid Tumors

STUDY DESIGN:
Intervention Model Description: 0.3mg/kg, 1.0mg/kg, 3.0mg/kg,10mg/kg，20mg/kg.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- XKH002 (Experimental): A total of 5 dose cohorts will be enrolled and treated: 0.3, 1.0, 3.0, 10, and 20 mg/kg. The dose-escalation process will utilize both the accelerated titration and the conventional 3+3 methods.
  Interventions: Drug: XKH002 Injection

INTERVENTIONS:
Drug: XKH002 Injection — 240 mg/4 mL/vial（60 mg/mL）
  Other Names: XKH002

SUMMARY:
This is a Phase 1, first-in-human (FIH), open-label, multicenter, dose-escalation and dose-expansion study to evaluate the safety, tolerability, pharmacokinetics, and antitumor activity of XKH002 in patients with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
Overall Study Design:

This is a Phase 1, first-in-human (FIH), open-label, multicenter, dose-escalation and dose-expansion study to evaluate the safety, tolerability, pharmacokinetics, and antitumor activity of XKH002 in patients with advanced or metastatic solid tumors.

The study will include 2 parts, dose escalation and dose expansion

Part 1: Dose Escalation Based on the results of previous non-clinical efficacy and toxicology experiments and the prediction of human PK, the initial dose was set at 0.3 mg/kg, and the dose was increased according to 5 dose groups: The 0.3, 1.0, 3.0, 10,20 mg/kg dose-escalation phase will include accelerated titration and a traditional 3+3 dose-escalation design, with 16-30 participants expected to participate in the study.

The MTD or MAD will be identified, and all the available PK, PD, tolerability and activity in addition to safety data will be evaluated to select the recommended dose for expansion (RDE).

Part 2: Dose Expansion Based on the results of the dose-escalation trial (safety/tolerability, initial efficacy, PK/PD, etc.), it is expected that 20 to 80 participants will be enrolled in the study by RDE dose expansion of monotherapy for selected subjects of 1 to 4 tumor types.

Number of Participants:

Approximately 16 to 30 patients will be enrolled in Part 1 (dose escalation). Approximately 20 to 80 patients will be enrolled in Part 2 (dose expansion).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. Life expectancy at least 3 months.
3. Histologically or cytologically confirmed unresectable locally advanced or metastatic solid tumor. Patient has had disease progression on one or more standard treatment regimens, or could not tolerate the treatment, or has no available treatment options.

4 The physical status score of "Eastern Cancer Collaboration Group (ECOG)" (see Appendix 5) was 0-1;

5 According to RECIST v1.1, all patients must have at least one evaluable lesion at baseline.

6 For patients with stable BMS, all of the following criteria must be met:

* At least 28 days after receiving specialist treatment for central nervous system disorders and at least 14 days after the last corticosteroid treatment.
* Clinical symptoms were stable after the last treatment: no new central nervous system metastases or radiotherapy complications.

Note: Patients who developed new progressive clinical symptoms or spinal cord compression or pIA disease after the last treatment were excluded.

7 Laboratory test results during the screening period meet all of the following criteria:

White blood cell count (WBC) ≥3.0×10^9/L;

* Neutrophil count (ANC) ≥1.5×10^9/L;
* Hemoglobin ≥90 g/L, assessed not having received blood transfusion within 7 days, and not dependent on erythropoietin (EPO);
* Platelets ≥90×10^9/L;
* Coagulation function: prothrombin time (PT), activated partial thromboplastin time (APTT), and International standardized ratio (INR) are all <1.5×ULN;
* No more than 1.5×ULN TBIL (no more than 3×ULN for Gilbert syndrome subjects);
* AST and/or ALT not higher than 3×ULN (or 5×ULN if liver metastasis is present);
* Albumin ≥30 g/L, no serum albumin infusion was assessed within 7 days;

Creatinine clearance (CrCl) ≥50 mL/min (calculated by Cockcroft-Gault formula).

8 Women with reproductive potential (refers to women who have not had birth control surgery and have been menopausal for less than 2 years) have negative serum pregnancy tests (human chorionic gonadotropin);

9 Fertile patients (men who have not had birth control, women who have not had birth control and have been menopausal for less than 2 years) must use a highly effective contraceptive method (such as oral contraceptives, intrauterine devices, abstinence or barrier contraception combined with spermicides) during the study and continue to use contraception for 6 months after the last dose;

10 Sign a written informed consent to participate in the study.

Exclusion Criteria:

1 The presence or history of any of the following:

Current or past autoimmune diseases or immunodeficiency, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener's granuloma, Sjogren's syndrome, Guillain-Barre syndrome, or multiple sclerosis, with the following exceptions (see Appendix 4) :

• Patients with autoimmune related hypothyroidism who only need thyroid hormone replacement therapy are eligible to participate in the study;

Patients with type 1 diabetes who receive insulin therapy for stable control are eligible to participate in the study;

Patients with only dermatologic clinical manifestations of eczema, psoriasis, chronic lichen simple or vitiligo (e.g., excluding psoriatic arthritis) are eligible to participate in the study if they meet all of the following criteria:

- The skin rash area must be < 10% of the body surface area;

* Good disease control at baseline, requiring only inefficient local glucocorticoid therapy;
* There has been no acute exacerbation of the pre-existing condition requiring psoralen plus A-band ultraviolet radiation, methotrexate, retinoic acid, biologics, oral calcineurin inhibitors, or highly effective or oral glucocorticoid therapy in the past 12 months.

  2.Known allergy to any component of XKH002;

  3 Subjects who had major surgery or were scheduled for surgery for any reason within the 4 weeks prior to screening or who the investigator felt might need surgery.

  4 Radiotherapy (except palliative radiotherapy), chemotherapy, targeted therapy, endocrine therapy and other anti-tumor therapy, or other clinical trial drugs should be administered within 4 weeks before the first dose to the end of the trial; a) Patients receiving oral fluorouracil or small molecule targeted drugs were discontinued for ≤2 weeks or 5 half-lives (whichever is longer) before the first administration of the drug in this study; b) Study patients who were treated with mitomycin C or nitrosourea within 6 weeks prior to first administration of the drug; c) Chinese medicines with anti-tumor indications should be used within 2 weeks before the first use of the investigational drug.

  5. Previous antibody/drug therapy targeting B7-H4 immune checkpoint;

  6 Pregnant or lactating women;

  7 Patients who have previously received allogeneic hematopoietic stem cell transplantation or solid organ transplantation;

  8 Patients receiving erythropoietin (EPO) or thrombopoietin (TPO) within 2 weeks before the first dose, or colony stimulating factor (CSF) within 1 week before the first dose;

  9 Confirmed by virological testing:

  • Active hepatitis B (HBsAg positive with HBV-DNA>500 IU/mL or lower limit of study center detection [only when lower limit of study center detection is higher than 500 IU/mL]), or

  • Active hepatitis C (patients with HCV antibody positive but HCV-RNA< lower limit of study center detection are allowed to be included), or

  • Known human immunodeficiency virus infection history or human immunodeficiency virus (HIV) antibody positive;

  10 ≥ grade 2 immune-related cardiotoxicity or ≥ grade 3 other immune-related adverse events after receiving immune checkpoint inhibitors or immune-modulating antibodies (immune-related hypothyroidism returning to grade 2 or below can be enrolled);

  11 has not recovered from the toxicity of previous systemic therapy, and still has NCI-CTCAE v5.0≥2 toxicity (except alopecia, platinum treatment-related neuropathy can be relaxed to grade 2);

  12 Concomitant diseases that may affect protocol adherence or interfere with trial results, including:

Cardiovascular disease: New York Heart Association (NYHA) Heart function Grade III or IV; Myocardial infarction, variable angina, or unstable angina in the past 6 months; Degree III atrioventricular block, malignant ventricular arrhythmias, and other potentially life-threatening arrhythmias within the past 6 months; Atrial fibrillation with uncontrolled ventricular rate;

* 12-lead ECG QTcF >470 ms for women and >450 ms for men;

Cardiac mural thrombosis, symptomatic deep vein thrombosis, and pulmonary embolism;

Note: Cardiac ultrasound is required in patients with a history of atrial fibrillation to exclude atrial mural thrombosis.

• Lung diseases: interstitial pneumonia, chronic obstructive pulmonary disease, active pulmonary tuberculosis and symptomatic bronchospasm;

Inflammatory gastrointestinal diseases, including Crohn's disease and ulcerative colitis;

* Chronic, active, clinically symptomatic infections, including bacterial, viral, fungal and other pathogens;
* Patients with severe complications such as active gastrointestinal bleeding, intestinal obstruction, intestinal paralysis, uncontrolled diabetes;
* Other severe and poorly managed comorbidities, in the opinion of the investigator.

  13 Receive live vaccine within 30 days before the first dose, or plan to receive live vaccine within 30 days of the first dose. Live vaccines include, but are not limited to, measles, mumps, rubella, varicella/shingles, rabies and typhoid vaccines. Allow seasonal influenza vaccine (usually inactivated);

  14 The novel coronavirus (COVID-19) vaccine is given within 14 days before the first dose, or is planned to be given within 14 days after the first dose, including the first dose, the second dose and the booster dose;

  15 A history of mental disorders, or a history of psychotropic drug and/or alcohol abuse that cannot be abated;

  16 Use immunosuppressive drugs. For corticosteroid users, systemic use of more than 10 mg/ day of prednisone or an equivalent dose of steroids must be discontinued at least 2 weeks before first administration of the test drug. Except in the following cases:
* Intranasal inhalation or local injection of corticosteroids;
* Continuous low dose (not exceeding 10 mg/d of prednisone or equivalent) for systemic use;

Short-term (no more than 3 days) systemic use of high-dose steroids (more than 10 mg/ day of prednisone or equivalent).

17 Patients with clinically uncontrollable third space effusion who were judged unsuitable for inclusion by the investigators;

18 The investigator considered that there were other reasons why the patient was not suitable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) or the maximum administered dose (MAD) and the recommended dose for expansion (RDE) | 24months
  To determine the maximum tolerated dose (MTD) or the maximum administered dose (MAD) and the recommended dose for expansion (RDE) of XKH002 in patients with advanced solid tumors
safety and tolerability | 24months
  Incidence of treatment emergent adverse events (TEAEs), abnormal clinical laboratory tests, vital signs, electrocardiogram (ECG), and physical examination

SECONDARY OUTCOMES:
pharmacokinetic (PK) parameters1 | 24months
  PK parameters including half-life (T1/2)
pharmacokinetic (PK) parameters2 | 24months
  PK parameters including clearance (CL)
pharmacokinetic (PK) parameters3 | 24months
  PK parameters including steady-state volume of distribution (Vss)
pharmacokinetic (PK) parameters4 | 24months
  PK parameters including area under the concentration-time (AUC)
pharmacokinetic (PK) parameters5 | 24months
  PK parameters including time to peak
pharmacokinetic (PK) parameters6 | 24months
  PK parameters including peak plasma concentration (Cmax)
antitumor activity1 | 24months
  To evaluate the antitumor activity of XKH002.Objective response rate (ORR)
antitumor activity2 | 24months
  To evaluate the antitumor activity of XKH002.disease control rate (DCR)
antitumor activity3 | 24months
  To evaluate the antitumor activity of XKH002. duration of overall response (DOR)
antitumor activity4 | 24months
  To evaluate the antitumor activity of XKH002.and progression-free survival (PFS)
antitumor activity5 | 24months
  To evaluate the antitumor activity of XKH002.according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)
immunogenicity | 24months
  To evaluate the immunogenicity of XKH002.Detection of antidrug antibodies (ADA)

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No